CLINICAL TRIAL: NCT01060163
Title: Effects of Antifibrinolytics on Bleeding and Transfusion Outcomes in Patients Receiving Coronary Artery Bypass Surgery With Preoperative Clopidogrel Exposure
Brief Title: Tranexamic Acid in Clopidogrel Exposure to Decrease Hemorrhage and Transfusion
Acronym: TRACED
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese Academy of Medical Sciences, Fuwai Hospital (Other)
Responsible Party: Principal Investigator, Li Lihuan, Professor and directior of the department of anaesthesiology, Cardiovascular Institute and Fuwai Hospital, Chinese Academy of Medical Sciences and Peking Union M, Chinese Academy of Medical Sciences, Fuwai Hospital
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Treatment
Other Study IDs: the TRACED trial
Record Dates: First submitted 2010-01-28; First posted 2010-02-02 (Estimated); Last update posted 2011-11-22 (Estimated); Status verified 2011-11

CONDITIONS: Coronary Artery Disease
Keywords: Clopidogrel; Tranexamic Acid; Cardiac Surgical Procedures; Hemostasis
MeSH Terms: conditions — Coronary Artery Disease | interventions — Tranexamic Acid; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (6):
- group ET (Experimental): Patients receiving early CABG <=7 days of the cessation of clopidogrel, treated with tranexamic acid with a bolus of 10 mg/kg after anesthetic induction and a maintenance of 10 mg/kg/h for the duration of surgery.
  Interventions: Drug: Tranexamic Acid
- group EP (Placebo Comparator): Patients receiving early CABG <= 7 days of the cessation of clopidogrel, treated with placebo(saline solution)
  Interventions: Drug: Saline
- group LT (Experimental): Patients receiving late CABG >7 days of the cessation of clopidogrel, treated with tranexamic acid with a bolus of 10 mg/kg after anesthetic induction and a maintenance of 10 mg/kg/h for the duration of surgery.
  Interventions: Drug: Tranexamic Acid
- group LP (Placebo Comparator): Patients receiving late CABG >7 days of the cessation of clopidogrel, treated with placebo(saline solution)
  Interventions: Drug: Saline
- group BT (Experimental): Patients receiving CABG without preoperative clopidogrel exposure, treated with tranexamic acid with a bolus of 10 mg/kg after anesthetic induction and a maintenance of 10 mg/kg/h for the duration of surgery.
  Interventions: Drug: Tranexamic Acid
- group BP (Placebo Comparator): Patients receiving CABG without preoperative clopidogrel exposure, treated with placebo(saline solution)
  Interventions: Drug: Saline

INTERVENTIONS:
Drug: Tranexamic Acid — A bolus of 10 mg/kg after anesthetic induction over 10 min followed by a maintenance of 10 mg/kg/h for the duration of surgery
  Arms: group BT; group ET; group LT
Drug: Saline — Saline served as placebo
  Arms: group BP; group EP; group LP

SUMMARY:
The use of platelet aggregation inhibitors, including aspirin and clopidogrel(CPDG), has become a standard management strategy for patients with acute coronary syndrome. On this background, an increasing percentage of patients presenting for surgical coronary revascularization is the subject to irreversible platelet inhibition.

Investigations on the effect of antiplatelet treatment on postoperative bleeding after cardiac surgery have shown that patients treated with antiplatelet agents until surgery have increased postoperative bleeding, and also an increased need for transfusions of blood products. As a result of the antiplatelet effect of clopidogrel, the frequency of serious bleeding complications has increased significantly, as seen in patients requiring coronary artery bypass grafting(CABG), especially when they received clopidogrel until surgery.

Tranexamic acid(TA) is a widely used antifibrinolytic agent, and is a promising substitute for aprotinin when the latter has seceded in 2007.The release of plasmin during cardiopulmonary bypass(CPB) activates fibrinolysis and may contribute to platelet dysfunction. Pharmacological inhibition of the fibrinolytic system may therefore ameliorate platelet dysfunction and fibrinolysis after CPB and decrease postoperative bleeding. Tranexamic acid prevents plasmin formation and inhibits fibrinolysis.

Concerning the cessation of aprotinin and the increasing proportion of patients with persistence on clopidogrel until their surgery, evolutional work is expected, especially in the eastern population.

The purpose of this study is to assess the effect of tranexamic acid in patients with clopidogrel and asprin ingestion until surgery. The investigators working hypothesis was that tranexamic acid would lower postoperative blood loss and transfusion requirements in these patients and would attenuate bleeding complication of antiplatelet therapy.

ELIGIBILITY:
Inclusion Criteria:

* Patients requiring primary and isolated coronary artery bypass grafting with cardiopulmonary bypass

Exclusion Criteria:

* history of cardiac surgery
* hematocrit <33%
* platelet count <100,000/ml
* allergy to tranexamic acid
* recruited in other studies

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 552 (Actual)
Dates: Start 2010-01; Primary Completion 2011-06 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
Postoperative blood loss(chest drainage) | on the 120th day postoperatively
Incidence of major bleeding | on the 120th day postoperatively
RBC Transfusion (volume and rate) | on the 120th day postoperatively

SECONDARY OUTCOMES:
Mortality | on the 120th day postoperatively
Major morbidity | on the 120th day postoperatively
  The major morbidity end points were defined as permanent disability caused by stroke, postoperative myocardial infarction, renal failure and respiratory failure.

CONTACTS AND LOCATIONS:
Overall Officials: Lihuang Li, MD, Study Chair — Cardiovascular Institute and Fuwai Hospital, CAMS&PUMC; Jia Shi, MD, Principal Investigator — Cardiovascular Institute and Fuwai Hospital, CAMS&PUMC
Locations (7):
- China (7):
  - Capital Medical University affiliated Beijing Anzhen Hospital, Beijing, Beijing Municipality
  - Cardiovascular Institute and Fuwai Hospital, CMAS&PUMC, Beijing, Beijing Municipality
  - General Hospital of Chinese People's Liberation Army, Beijing, Beijing Municipality
  - Fujian Provincial Hospital, Fuzhou, Fujian
  - Shanghai Jiaotong University affiliated Chest Hospital, Shanghai, Shanghai Municipality
  - the Fourth Military Medical University affiliated Xijing Hospital, Xi’an, Shanxi
  - TEDA International Cardiovascular Hospital, Tianjin, Tianjin Municipality

REFERENCES:
- [Derived] Shi J, Ji H, Ren F, Wang G, Xu M, Xue Y, Chen M, Qi J, Li L. Protective effects of tranexamic acid on clopidogrel before coronary artery bypass grafting: a multicenter randomized trial. JAMA Surg. 2013 Jun;148(6):538-47. doi: 10.1001/jamasurg.2013.1560. PMID 23426385